CLINICAL TRIAL: NCT04630873
Title: Different Dilutions and Efficacy of Botulin Toxin in the Correction of the Hemiplegic Gait
Brief Title: Low or High Botox Dilution for the Hemiplegic Gait?
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Ioannina (Other)
Responsible Party: Principal Investigator, Avraam Ploumis, Professor of Physical Medicine and Rehabilitation, University of Ioannina
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: UIoannina 2
Record Dates: First submitted 2020-10-31; First posted 2020-11-16 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Post Stroke Spastic Hemiplegia
Keywords: stroke; hemiplegia
MeSH Terms: conditions — Stroke; Hemiplegia | interventions — Botulinum Toxins; Gait Analysis

STUDY DESIGN:
Intervention Model Description: In a sequential manner, every second patient that will meet our inclusion criteria will be treated with a low concentration of the drug during their first visit at our outpatient clinic. Then, after a safe washout period of 6 months, the same patients will be injected with a high concentration of the drug. The same procedure will be inversely performed in the other half of the patients.
Who Masked: Care Provider, Investigator
Masking Description: In a sequential manner, every second patient that will enter the protocol will be treated with one of the two (high or low) diluted drug and will be assigned a number. Neither the investigator nor the outcome assessor (who will read the gait parameters) will be aware of the dilution used in each case.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- LOW-HIGH VOLUME (Active Comparator): Initially a low volume of the drug (100IU botulinum toxin diluted in 2 ml) after a safe washout period of 6 months the same patients will be injected with a high volume (100IU botulinum toxin in 4 ml) of the drug.
  Interventions: Drug: Botulinum toxin; Diagnostic Test: gait analysis
- HIGH-LOW VOLUME (Experimental): initially a high volume of the drug (100IU botulinum toxin diluted in 4 ml) after a safe washout period of 6 months the same patients will be injected with a low volume (100IU botulinum toxin in 2 ml) of the drug.
  Interventions: Drug: Botulinum toxin; Diagnostic Test: gait analysis

INTERVENTIONS:
Drug: Botulinum toxin — The triceps surae along with the posterior tibialis muscle will be injected. The units that will be injected are the average being injected in our University Clinic. I.e. 50 units for each head of the gastrocnemius muscle- single injection site, 100 units for the soleus muscle- two injection sites and 50 units for the posterior tibialis muscle- single injection site.
Diagnostic Test: gait analysis — The gait analysis will be performed with two systems. A foot pressure sensitivity walkway (medicapteurs Win-Track), and an IMU network system (RehaGait Pro) using seven IMU's placed in specific anatomical positions. In combination those two systems can provide a wide range of spatiotemporal analytics of gait:
  Other Names: medicapteurs Win-Track; RehaGait Pro

SUMMARY:
There is debate regarding the efficiency of different dilutions of Botulin toxin type A (BTX-A) injections. Some authors believe that highly diluted BTX-A injections achieve greater neuromuscular blockade resulting in higher spasticity reduction. On the other hand, other researchers suggest that there is no difference in spasticity decrease if either high or low volume toxin is being injected. Studies on this subject lack either the design or the power of study was low. Therefore, there is no clear guideline for an optimal botulinum toxin dilution protocol. In an attempt to have a better understanding, a cross over study was designed. The material will be patients with spastic hemiparesis which will be treated with Botulin toxin at different dilutions. Gait analysis will be used for the evaluation of the Botulin toxin injection on gait improvement. To the best of our knowledge such a trial hasn't been performed yet.

DETAILED DESCRIPTION:
There is an ongoing controversy regarding the effect of different dilutions in the efficacy of Botulin toxin type A (BTX-A) injections. Some authors believe that highly diluted BTX-A injections achieve greater neuromuscular blockade resulting in higher spasticity reduction. They are arguing that BTX-A in high dilution is the optimal choice especially when bigger muscles are injected, for the large volume of fluid administered into the muscle will carry the BTX-A molecules to endplates remote from the injection site. Two animal studies suggest that increasing the volume of diluents is a potential strategy in order to achieve a more efficient and cost-effective manner of BTX-A treatment. An attempt to quantify how the location of BTX-A injection affects the drug effect was made, which revealed that injecting only 0.5 cm away from the motor endplates yielded a 50% decrease in paralysis2. A newer double-blinded study by JM Gracies et al performed on humans comes to the same conclusion, that high volume dilution provides greater neuromuscular block and spasticity reduction than a low volume dilution. On the other hand, other researchers suggest that there is no difference in spasticity decrease if either high or low volume toxin is being injected.

Previous studies lack either the design or the power of study was low. Therefore, there is no clear guideline for an optimal botulinum toxin dilution protocol.

ELIGIBILITY:
Inclusion Criteria:

* equinovarus deformity
* with an average 3 on Ashworth spasticity scale
* able to walk indoors either freely or with a cane.

Exclusion Criteria:

* patients suffering from any mental illness that would disturb the gait pattern
* patients suffering from musculoskeletal diseases that overtly interfere with the gait

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-11-20 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Change of Ankle motion from baseline to 1 month postinjection | Day 1 (baseline) and at 1 month postinjection
  range of motion of ankle during gait
Change of modifies Ashworth scale (from 0 to 4, higher grade means worse spasticity) of the ankle from baseline to 1 month postinjection | Day 1 (baseline) and at 1 month postinjection
  spasticity measurement
Change of standing balance from baseline to 1 month postinjection | Day 1 (baseline) and at 1 month postinjection
  measuring the ground force position when standing
Change of walking balance from baseline to 1 month postinjection | Day 1 (baseline) and at 1 month postinjection
  measuring the ground force position when walking

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Medicine and Rehabilitation, University Hospital of Ioannina, Ioannina, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Francisco GE, Boake C, Vaughn A. Botulinum toxin in upper limb spasticity after acquired brain injury: a randomized trial comparing dilution techniques. Am J Phys Med Rehabil. 2002 May;81(5):355-63. doi: 10.1097/00002060-200205000-00007. PMID 11964576
- [Background] Lee LR, Chuang YC, Yang BJ, Hsu MJ, Liu YH. Botulinum toxin for lower limb spasticity in children with cerebral palsy: a single-blinded trial comparing dilution techniques. Am J Phys Med Rehabil. 2004 Oct;83(10):766-73. doi: 10.1097/01.phm.0000137314.38806.95. PMID 15385785
- [Result] Gracies JM, Lugassy M, Weisz DJ, Vecchio M, Flanagan S, Simpson DM. Botulinum toxin dilution and endplate targeting in spasticity: a double-blind controlled study. Arch Phys Med Rehabil. 2009 Jan;90(1):9-16.e2. doi: 10.1016/j.apmr.2008.04.030. PMID 19154823
- [Result] Shaari CM, Sanders I. Quantifying how location and dose of botulinum toxin injections affect muscle paralysis. Muscle Nerve. 1993 Sep;16(9):964-9. doi: 10.1002/mus.880160913. PMID 8355728
- [Result] Pearce LB, Borodic GE, First ER, MacCallum RD. Measurement of botulinum toxin activity: evaluation of the lethality assay. Toxicol Appl Pharmacol. 1994 Sep;128(1):69-77. doi: 10.1006/taap.1994.1181. PMID 8079356